CLINICAL TRIAL: NCT04038346
Title: Symptomatic Management of Lyme Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study with overlapping patient population
Sponsor: Desiree Neville, MD (Other)
Responsible Party: Sponsor-Investigator, Desiree Neville, MD, Assistant Professor of Pediatric Emergency Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20040185
Record Dates: First submitted 2019-07-15; First posted 2019-07-30 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Lyme Arthritis; Lyme Disease; Arthritis
Keywords: Lyme Arthritis; Lyme; Lyme Disease; Arthritis; NSAID
MeSH Terms: conditions — Lyme Disease; Arthritis | interventions — Naproxen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, non blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- NSAID (Experimental): Naproxen at weight based standard dose given bid daily until symptoms resolve
  Interventions: Drug: Naproxen
- Acetaminophen (Active Comparator): Acetaminophen at weight based standard dose given qid until symptoms resolve
  Interventions: Drug: Acetaminophen
- NSAID first, then Acetaminophen (Experimental): Naproxen at weight based standard dose given bid for one week, then acetaminophen at weight based standard dose given qid until symptoms resolve
  Interventions: Drug: Naproxen; Drug: Acetaminophen
- Standard Care (No Intervention): Symptom observation only

INTERVENTIONS:
Drug: Naproxen — Patients will be randomized to an NSAID (naproxen)
  Other Names: naprosyn, aleve, anaprox
  Arms: NSAID; NSAID first, then Acetaminophen
Drug: Acetaminophen — Patients will be randomized to acetaminophen
  Other Names: tylenol
  Arms: Acetaminophen; NSAID first, then Acetaminophen

SUMMARY:
Lyme arthritis resolves with appropriate antimicrobial treatment in a majority of patients, but 10-20% of patients develop antibiotic-refractory Lyme arthritis with prolonged arthritis symptoms and treatment courses. Excessive up-regulation of the inflammatory process has been shown in patients with antibiotic-refractory Lyme arthritis. The over-expressed pro-inflammatory cell mediators are downstream of NSAID inhibition, which would suggest initial inflammatory inhibition may be beneficial in these patients. While NSAIDs are known to reduce pro-inflammatory cell mediators early in the course of inflammation, research has shown that there are other cytokines that play a role in the healing after inflammation that are also inhibited by NSAIDs, and that NSAID use can delay healing.

It is not known if scheduled NSAID therapy will reduce, increase, or have no effect on the occurrence of refractory Lyme arthritis cases. The hypothesis of the study is that prescribing scheduled NSAIDs at the time of diagnosis of Lyme arthritis can prevent the development of the excessive inflammatory phase and decrease the number of patients with antibiotic-refractory Lyme arthritis, or at least decrease the duration of persistent Lyme arthritis symptoms.

The pilot study design randomizes patients to scheduled NSAIDs, scheduled acetaminophen, or scheduled NSAIDs x 1 week than acetaminophen. Primary outcomes are duration of arthritis symptoms, number of refractory cases, side effects and compliance.

DETAILED DESCRIPTION:
Specific Aims:

1. Demonstrate feasibility to ensure adequate patient enrollment and symptomatic follow-up of patients with Lyme arthritis.
2. Develop pilot data necessary for sample size and power calculations:

The purpose of the research study is to evaluate whether there is symptomatic benefit of schedule NSAID therapy in patients with Lyme arthritis diagnosis.

1. Quantification of antibiotic-refractory Lyme arthritis in our population
2. Symptomatic outcomes of patients with Lyme arthritis on scheduled NSAIDs versus those not placed on scheduled NSAIDs (duration to resolution and number of patients with resistant arthritis)
3. Assess side effects of patients with Lyme arthritis placed on scheduled NSAIDs versus those not placed on scheduled NSAIDs
4. Assess changes in resources (follow-up visits, further prescriptions) required for patients taking scheduled NSAIDs versus not taking scheduled NSAIDs

Background:

Lyme disease is the systemic tick-borne disease caused by Borrelia burgdorferi infection, and is endemic to an expanding portion of the United States. Lyme arthritis is a common presentation of Lyme disease. While Lyme arthritis resolves with appropriate antimicrobial treatment in a majority of patients, 10-20% of patients develop antibiotic-refractory Lyme arthritis with prolonged inflammatory arthritis. Research suggests excessive up-regulation of the inflammatory process in patients with prolonged symptoms. The over-expressed pro- inflammatory cell mediators are downstream of NSAID inhibition, which would suggest NSAIDs may be beneficial in these patients. In fact, there is data that NSAIDs and/or disease-modifying anti-rheumatic drugs (DMARDs) may be beneficial in refractory Lyme arthritis cases, once diagnosed as refractory.

The hypothesis of the study is that prescribing scheduled NSAIDs at the time of diagnosis can prevent the development of the excessive inflammatory phase and decrease the number of patients with antibiotic-refractory Lyme arthritis, or at least decrease the duration of persistent Lyme arthritis symptoms. There are no known methods to identify patients who will develop antibiotic-refractory Lyme arthritis. This work is important to delineate optimal timing and duration of NSAIDs given the research that shows the anti- inflammatory effects during healing can potentially delay recovery.

Significance:

While antibiotic-refractory Lyme arthritis has been studied at a microbiologic/cytokine level as well as evaluated in terms of treatment once patients have been deemed antibiotic refractory, to our knowledge there are no published studies evaluating prevention.

With no literature looking at the question of NSAIDs for the prevention of antibiotic- refractory Lyme arthritis, this pilot study is needed to adequately calculate sample size and power calculations for a large-scale multicenter study. There is anecdotal data from the Rheumatology and Infectious Disease departments at the UPMC Children's Hospital of Pittsburgh that early scheduled NSAIDs may decrease refractory cases, but there has been no formal evaluation into this question. Retrospective evaluation is challenging since the medications in question (NSAIDs) are over the counter, and clinicians may recommend scheduled or intermittent NSAID therapy without documentation, and certainly without prescriptions in the medical record. Many patients with refractory Lyme arthritis are placed on NSAIDs, but given the question of delayed healing with inhibition of prostaglandins during the healing phase of inflammation, the question of whether NSAIDs are beneficial in patients to prevent refractory arthritis is worthwhile rather than the current process of variable NSAID prescription.

ELIGIBILITY:
Inclusion Criteria:

* Arthritis
* Undergoing Lyme disease testing (Lyme test positive)

Exclusion Criteria:

* Patients will be secondarily withdrawn from analysis and instructed to stop study medication if their Lyme test is negative.

Underlying diagnosis of rheumatoid or recurrent arthritis Already on scheduled NSAIDs

Anything that restricts the prescription of naproxen or acetaminophen:

* Hypersensitivity to naproxen (for example: anaphylactic reactions, serious skin reactions) or any component of the formulation; history of aspirin induced asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs, underlying kidney or liver impairment
* Already taking daily NSAIDs (naproxen or ibuprofen) or daily acetaminophen
* Hypersensitivity to acetaminophen or any component of the formulation; severe liver impairment or severe active liver disease

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desiree NW Neville, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Started | 1 | 2 | 0 | 0
Completed | 1 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 3 patients were enrolled in two arms before enrollment pause.
Groups:
- Total: Total of all reporting groups
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care | Total
Number analyzed (Participants) | 1 | 2 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 0 | 0 | 3
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 9 [9 to 9] | 6 [6 to 6] |  |  | 7 [6 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 |  |  | 2
  Male | 0 | 1 |  |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Joint Pain Reported by Serial Visual Analog Scale (VAS) for Pain Via Text Surveys
Description: 0-100 scale (no pain to worst pain - higher score, worse outcome), slide bar in text survey
Time Frame: days 0(enrollment), 1, 3, 7, 10, 14, 21, 28, 60 the VAS score will be collected
Population: VAS score for pain across all groups
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
score on a scale
  Enrollment, Day 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Enrollment, Day 0 | 62 [62 to 62] | 58 [58 to 58] |  |
  Day 1 | 50 [50 to 50] | 49.5 [49 to 50] |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 16 [16 to 16] | 26 [26 to 26] |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 0 [0 to 0] |  |  |
  Day 10: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 10 | 0 [0 to 0] |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 20 [20 to 20] |  |
  Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 21 | 0 [0 to 0] |  |  |
  Day 28: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 28 | 0 [0 to 0] |  |  |
  Day 60: number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Joint Redness Reported by Serial Visual Analog Scale for Joint Redness Via Text Surveys
Description: 0-100 scale (no redness to maximal redness- higher score, worse outcome), slide bar in text survey
Time Frame: days 0 (enrollment), 1, 3, 7, 10, 14, 21, 28, 60 the VAS score for join redness will be collected
Population: There was not 100% follow-up with text surveys
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
score on a scale
  Enrollment, Day 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Enrollment, Day 0 | 61 [61 to 61] | 20 [20 to 20] |  |
  Day 1 | 38 [38 to 38] | 22.5 [12 to 33] |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 7 [7 to 7] | 19 [19 to 19] |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 0 [0 to 0] |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 0 [0 to 0] |  |
  Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 21 | 0 [0 to 0] |  |  |
  Day 28: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 28 | 0 [0 to 0] |  |  |
  Day 60: number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Joint Movement Reported by Serial Visual Analog Scale for Joint Movement Via Text Surveys
Description: 0-100 scale (no joint movement to normal joint movement- higher score, better outcome), slide bar in text survey
Time Frame: days 0 (enrollment), 1, 3, 7, 10, 14, 21, 28, 60 the VAS score for joint movement will be collected
Population: Not all text survey instances completed.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
score on a scale
  Enrollment, Day 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Enrollment, Day 0 | 35 [35 to 35] | 50 [50 to 50] |  |
  Day 1 | 50 [50 to 50] | 47 [37 to 57] |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 86 [86 to 86] | 78 [78 to 78] |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 100 [100 to 100] |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 84 [84 to 84] |  |
  Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 21 | 100 [100 to 100] |  |  |
  Day 28: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 28 | 100 [100 to 100] |  |  |
  Day 60: number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Overall Function Reported by Serial Visual Analog Scale for Overall Function Via Text Surveys
Description: 0-100 scale (severely impaired function to normal function- higher score, better outcome), slide bar in text survey
Time Frame: days 0 (enrollment), 1, 3, 7, 10, 14, 21, 28, 60 the VAS score will be collected
Population: Not all text surveys completed.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
score on a scale
  Enrollment, Day 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Enrollment, Day 0 | 50 [50 to 50] | 50 [50 to 50] |  |
  Day 1 | 65 [65 to 65] | 55.5 [50 to 61] |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 85 [85 to 85] | 89 [89 to 89] |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 100 [100 to 100] |  |  |
  Day 10: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 10 | 100 [100 to 100] |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 83 [83 to 83] |  |
  Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 21 | 100 [100 to 100] |  |  |
  Day 28: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 28 | 100 [100 to 100] |  |  |
  Day 60: number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Time to Complete Symptom Resolution as Collected by a Yes/no Question on the Text Survey
Description: If patient answers yes to symptoms completely resolved, the time frame from enrollment will be the days to symptom resolution
Time Frame: Symptom resolution recorded (days 0, 1, 3, 7, 10, 14, 21, 28, 60) once they enter "yes" to symptoms completely resolved
Population: 3 enrolled patients - none of the acetaminophen patients continued until resolution
Measure: Mean (Full Range); unit: days since enrollment
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 0 | 0 | 0
days since enrollment | 6 [6 to 6] |  |  |

6. Secondary Outcome: Medication Compliance as Determined by Question in Serial Text Survey
Description: Parents enter number of days patient has taken the medication in the past day as well as per day since the last survey in two questions on the text survey with their response being a drop down number list on the text survey- medication compliance will be compared to the number of doses that would be full compliance for that treatment arm
Time Frame: days 1, 3, 7, 10, 14, 21, 28, 60 (collected until symptom resolution)
Population: Randomized participants, report percentage of medication doses taken that were available. (while still reporting symptoms)
Measure: Mean (Full Range); unit: percentage of available med doses taken
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
percentage of available med doses taken
  Day 1 | 100 [100 to 100] | 75 [75 to 75] |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 100 [100 to 100] | 100 [100 to 100] |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 100 [100 to 100] |  |  |
  Day 10: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 10 | 100 [100 to 100] |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 25 [25 to 25] |  |
  Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 28: number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: The Number of Participants With Reported Medication Side Effects as Determined by Question in Serial Text Survey
Description: survey asks parents to describe any medication side effects they feel their child has had - descriptive outcome only
Time Frame: days 1, 3, 7, 10, 14, 21, 28, 60 (collected until symptom resolution)
Population: Randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
Participants
  Day 1 | 0 | 0 |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 0 | 0 |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 1 |  |  |
  Day 10: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 10 | 0 |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 0 |  |
  Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 21 | 0 |  |  |
  Day 28: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 28 | 0 |  |  |

8. Secondary Outcome: The Number of Participants Who Reported Taking Other Medications as Determined by Question in Serial Text Survey
Description: Parents are asked to list any medications in addition to their study drug and the prescribed antibiotic that their child has taken- descriptive outcome only
Time Frame: days 1, 3, 7, 10, 14, 21, 28, 60 (collected until symptom resolution)
Population: randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
Participants
  Day 1 | 0 | 0 |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 0 | 0 |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 0 |  |  |
  Day 10: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 10 | 0 |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 0 |  |
  Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 21 | 0 |  |  |
  Day 28: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 28 | 0 |  |  |
  Day 60: number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Reported Fever as Determined by Question in Serial Text Survey
Description: Parents are asked if their child had fever in the 24 hours prior to taking the text survey
Time Frame: days 0 (enrollment), 1, 3, 7, 10, 14, 21, 28, 60 (collected until symptom resolution)
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
Participants
  Day 0 (Enrollment): number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 0 (Enrollment) | 1 | 0 |  |
  Day 1 | 0 | 1 |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 3 | 0 | 0 |  |
  Day 7: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 7 | 0 |  |  |
  Day 10: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 10 | 0 |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 14 |  | 0 |  |
  Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 21 | 0 |  |  |
  Day 28: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 28 | 0 |  |  |

10. Other Pre Specified Outcome: Need for Further Care as Determined by Medical Record Review as Mean Number of Visits in the System for Lyme Arthritis Symptoms During Each Time Frame
Description: Mean repeat medical visits for Lyme arthritis will be compared between treatment arms based on medical record review
Time Frame: 30 days, 60 days, 120 days, 1 year
Population: All patients were analyzed for return visits by: 30 days, 60 days, 120 days, 1 year
Measure: Mean (Full Range); unit: return visits for Lyme arthritis symptom
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
Number analyzed (Participants) | 1 | 2 | 0 | 0
return visits for Lyme arthritis symptom
  30 days | 0 [0 to 0] | 0 [0 to 0] |  |
  60 days | 0 [0 to 0] | 0 [0 to 0] |  |
  120 days | 0 [0 to 0] | 0 [0 to 0] |  |
  1 year | 0 [0 to 0] | 0 [0 to 0] |  |

ADVERSE EVENTS:
Time Frame: Collected by text surveys at days from enrollment: 0, 1, 3, 7, 10, 14, 21, 28, 60 until asymptomatic.
Description: Collected by text surveys at days from enrollment: 0, 1, 3, 7, 10, 14, 21, 28, 60. Question: Have you noticed any medication side-effects.
Arm/Group | NSAID | Acetaminophen | NSAID First, Then Acetaminophen | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/2 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSAID (N=1) | Acetaminophen (N=2) | NSAID First, Then Acetaminophen (N=0) | Standard Care (N=0)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — one episode of emesis reported on day 7 survey

LIMITATIONS AND CAVEATS:
The study was stopped prematurely due to Covid research pause and then overlapping study populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT04038346/Prot_001.pdf